CLINICAL TRIAL: NCT02247609
Title: Safety and Efficacy Evaluation of 4th Generation Safety-engineered CAR T Cells Targeting High-risk and Refractory B Cell Lymphomas
Brief Title: Evaluation of 4th Generation Safety-designed CAR T Cells Targeting High-risk and Refractory B Cell Lymphomas
Acronym: 4SCAR19273
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19273-4SCAR
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-01

CONDITIONS: B-cell Lymphomas
Keywords: B cell lymphoma; non-Hodgkin's lymphoma; Burkitt lymphoma; diffused large B cell lymphoma; B cell malignancy
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR T cells (Experimental): Autologous 4th generation anti-CD19-CAR T cells
  Interventions: Genetic: Anti-CD19 CAR T cells

INTERVENTIONS:
Genetic: Anti-CD19 CAR T cells — Autologous 4th generation withdrawable lentiviral-transduced anti-CD19-CAR T cells
  Other Names: 19273-4SCAR

SUMMARY:
Currently, a majority of B cell lymphomas cannot be cured by standard chemo-radiotherapy. Most B cell lymphomas express cluster of differentiation antigen 19 (CD19), which represents a very attractive target for chimeric antigen receptor (CAR)-based immune cell therapy. This study will evaluate a novel 4th generation CD19 CAR engineered with a self-withdrawal mechanism (19273-4SCAR) for both efficacy and safety in lymphoma patients.

DETAILED DESCRIPTION:
CD19 single chain antibody-based chimeric antigen receptor (CAR)-engineered T cells have demonstrated great clinical potential in treating chronic and acute B cell leukemias. B cell lymphomas, similar to B cell leukemias, express CD19 surface molecules, and the majority of the B cell lymphoma patients cannot be cured by standard chemo-radiotherapy. CD19 CAR-based adoptive T cell therapy is associated with an unwanted adverse effect, the loss of CD19 B cells, which results in humoral immune deficiency. This study will evaluate a novel 4th generation CD19 CAR engineered with a self-withdrawal genetic mechanism (19273-4SCAR) for both efficacy and safety in lymphoma patients. The 4th generation design of the CAR incorporates the intracellular signaling domain of cluster of differentiation antigen 27 (CD27), known to be associated with T cell activation, survival and longevity. The inducible caspase 9 self-withdrawal design allows for rapid elimination of the infused CAR T cells upon complete eradication of the tumor cells, which will be followed by the recovery of humoral immunity. Patients receiving the 19273-4SCAR T cells will be closely monitored for infusion response, tumor eradication effect, longevity of the CAR T cells, and the recovery of B cell functions after withdrawal of the CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD19(+) B cell lymphoma patients proved by immuno-histochemistry (IHC) or Flow-cytometry.
* Not eligible for autologous stem-cell transplantation (ASCT) or relapsed after ASCT.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Age≥18.
* Pulse oximetry of > 90% on room air.
* Adequate hepatic function, defined as alanine transaminase (ALT) <3 x upper limit of normal (ULN), aspartate aminotransferase (AST) <3 x ULN; serum bilirubin and alkaline phosphatase <2 x ULN.
* Adequate renal function, defined as serum creatinine <2.0mg/dl.
* Adequate heart function with LVEF≥50%
* Hb≥80g/L
* Measurable disease can be identified.
* Life expectancy ≥3 months.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 1 year after the study is concluded. The male partner should use a condom.
* Patients must sign an informed consent.

Exclusion Criteria:

* Uncontrolled active infection.
* Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV).
* HIV positive
* Pregnant or lactating.
* Currently enrolled in another clinical trial.
* Concurrent use of systemic steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 2 years.
  Determine the toxicity profile of the 4th generation CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-CD19 CAR T cells in vivo. | 2 years.
  Measure the survival of 4th generation CAR T cells transduced with the anti-CD19 lentiviral vector.
Response rates to the 4th generation CAR T cells. | 2 years.
  Describe the response rates of patients treated with 4th generation CAR T cells, including partial remission (PR), complete remission (CR), stable disease (SD) and progressive disease (PD).
Survival time of the patients. | 2 years.
  Evaluate the survival time of the patients treated with the 4th generation CAR T cells, including progression free survival (PFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China